CLINICAL TRIAL: NCT00144521
Title: A Double-Blind, Phase III Study to Evaluate the Efficacy and Safety of MRA in Patients With RA
Brief Title: Comparative Study (Double-Blind) of MRA for Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRA213JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MRA(Tocilizumab); Drug: MTX placebo
- 2 (Active Comparator)
  Interventions: Drug: MRA placebo; Drug: MTX

INTERVENTIONS:
Drug: MRA(Tocilizumab) — 8mg/kg/4week(i.v.)for 24 weeks
  Arms: 1
Drug: MRA placebo — 0mg/kg/4week(i.v.) for 24 weeks
  Arms: 2
Drug: MTX — 8mg/week(p.o.) for 24 weeks
  Arms: 2
Drug: MTX placebo — 0mg/week(p.o.) for 24 weeks
  Arms: 1

SUMMARY:
The purpose of this study is to investigate the clinical efficacy and safety of MRA in a double-blind, parallel-group, controlled study using MRA or methotrexate (MTX) in rheumatoid arthritis (RA) patients with MTX administered.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of RA based on the 1987 classification criteria of the American College of Rheumatology (ACR)
* Disease duration of 6 months or more
* Treated with 8 mg/week of MTX for at least 8 weeks immediately preceding enrollment, and continued on this treatment up to initiation of the study drug
* Active disease at enrollment (less than 2 weeks before initiating treatment with a study drug), Which is defined as having at least 6 tender and 6 swollen joints among 49 and 46 joints stipulated by the Japanese Rheumatism Foundation's Drug Evaluation Committee and ESR at least 30 mm/hr and CRP not less than 1.0 mg/dL

Exclusion criteria

* Assessed as having Class IV Steinbrocker functional activity in the 4 weeks preceding treatment with the study drug
* Treated with infliximab, etanercept or leflunomide in the 12 weeks preceding treatment with the study drug
* Received any of the following therapies in the 2 weeks preceding initiation of treatment with the study drug.

  1. Administration of any DMARD or immunosuppressant other than MTX
  2. Administration of corticosteroids exceeding 10 mg/day as prednisolone
  3. Dose escalation or initiation of corticosteroids
* Received any of the following therapies in the 4 weeks preceding treatment with the study drug

  1. Plasma exchange therapy
  2. Surgical treatment (operation, etc.)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2004-02; Primary Completion 2004-08 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Frequency of ACR 20% improvement | week 24

SECONDARY OUTCOMES:
Frequency and severity of adverse events and adverse drug reactions | throughout study
Time course of DAS28 | throughout study
time course of the frequency of ACR 20%, 50% and 70% | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical